CLINICAL TRIAL: NCT01263093
Title: Effect of LY2216684 on the Pharmacokinetics and Pharmacodynamics of R-130964, the Active Metabolite of Clopidogrel, in Healthy Subjects
Brief Title: A Pharmacokinetic Study on the Effect of LY2216684 on the Active Metabolite of Clopidogrel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12593; H9P-EW-LNBY (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Clopidogrel; alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel First, Then LY2216684 + Clopidogrel (Experimental): Period 1: a single 300-milligram (mg) dose of clopidogrel administered orally on Day 1 (Treatment 1).
  Period 2: an 18-mg dose of LY2216684 administered orally, once daily (QD) on Days 1 through 3, plus a single 300-mg dose of clopidogrel administered orally on Day 3 (Treatment 2).
  There was a washout period of at least 14 days between the last dose of study drug in Period 1 and the first dose in Period 2.
  Interventions: Drug: Clopidogrel; Drug: LY2216684
- LY2216684 + Clopidogrel First, Then Clopidogrel (Experimental): Period 1: an 18-milligram (mg) dose of LY2216684 administered orally, once daily (QD) on Days 1 through 3, plus a single 300-mg dose of clopidogrel administered orally on Day 3 (Treatment 2).
  Period 2: a single 300-mg dose of clopidogrel administered orally on Day 1 (Treatment 1).
  There was a washout period of at least 14 days between the last dose of study drug in Period 1 and the first dose in Period 2.
  Interventions: Drug: Clopidogrel; Drug: LY2216684

INTERVENTIONS:
Drug: Clopidogrel
Drug: LY2216684

SUMMARY:
The purpose of this study is to measure how much of the study drugs (clopidogrel and LY2216684) reach the blood stream and how long it takes the body to dispose of them and to determine how clopidogrel and LY2216684 might affect each other in the body. Information about any side effects that may occur will also be collected.

DETAILED DESCRIPTION:
Clopidogrel is rapidly converted to R-130964 by the enzyme cytochrome P450 2C19 (CYP2C19). Enrollment in the study was limited to participants with specific genotypes of the CYP2C19 gene, including the *1/*1 genotype (CYP2C19 extensive metabolizers) and the *1/*17 or *17/*17 genotypes (CYP2C19 ultra-rapid metabolizers). All primary and secondary objectives were limited to participants with the CYP2C19*1/*1 genotype.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy, as determined by medical history and physical examination.
* Male participants - Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug.
* Female participants - Women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone [FSH] >40 milli-international units per milliliter [mIU/mL]).
* Have a body weight >50 kilograms (kg).
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow blood sampling as per the protocol.
* Have normal blood pressure and pulse rate (sitting position) as determined by the investigator.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site.
* Are cytochrome P450 (CYP) 2C19 extensive metabolizers or ultra -rapid metabolizers as determined by genotyping assessment.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device other than the study drug, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to LY2216684, clopidogrel, or related compounds.
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to screening.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have a history of or show evidence of significant active neuropsychiatric disease or have a history of suicide attempt or ideation.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing unless deemed acceptable by the investigator and Sponsor's medical monitor, except for influenza vaccinations.
* Use of any drugs or substances that are known to be substrates, inducers, or inhibitors of CYP2C19 or CYP3A4 within 30 days prior to dosing.
* Have donated blood of more than 500 milliliters (mL) within the last month.
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption 48 hours prior to check-in until completion of the study (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any participants unwilling to adhere to study caffeine restrictions.
* Have used any tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to enrollment.
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment and during the study.
* Have a documented or suspected history of glaucoma.
* History or presence of significant bleeding disorders that is, haematemesis, melanena, severe or recurrent epistaxis, haemoptysis, clinically overt clinical haematuria or intracranial haemorrhage.
* Participants with a history of gastrointestinal ulcers or haemorrhage.
* Personal or family history of coagulation or bleeding disorders or reasonable suspicion of vascular malformations, for example, cerebral haemorrhage, aneurysm or premature stroke (cerebrovascular accident <65 years of age).
* Self-reported history of increased bleeding from trauma (for example, prolonged bleeding after tooth extraction).
* History of major surgery within 3 months of screening.
* Planned surgery within 14 days after the last day of dosing.
* International normalized ratio (INR), prothrombin time (PT), activated partial thromboplastin time (APTT) above the normal reference range or platelet count below the normal reference range at screening.
* Positive fecal occult blood examination at screening.
* Clinically significant abnormality in fundoscopic or petechiae examination.
* Consumption of aspirin, other non-steroidal anti-inflammatory drugs or other drugs known to affect platelet function within 21 days prior to dosing.
* Participants determined to be unsuitable by the investigator for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Clopidogrel First, Then LY2216684 + Clopidogrel | LY2216684 + Clopidogrel First, Then Clopidogrel
Started | 24 | 23
Completed | 24 | 23
Not Completed | 0 | 0
Period: Washout
Arm/Group | Clopidogrel First, Then LY2216684 + Clopidogrel | LY2216684 + Clopidogrel First, Then Clopidogrel
Started | 24 | 23
Completed | 23 | 23
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Period 2
Arm/Group | Clopidogrel First, Then LY2216684 + Clopidogrel | LY2216684 + Clopidogrel First, Then Clopidogrel
Started | 23 | 23
Completed | 22 | 23
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel First, Then LY2216684 + Clopidogrel | LY2216684 + Clopidogrel First, Then Clopidogrel | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (11.2) | 44.5 (11.5) | 42.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 12 | 28
  Not Hispanic or Latino | 8 | 11 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of R-130964, Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-∞)
Description: R-130964 is the active metabolite of clopidogrel. Blood samples were collected prior to and through 24 hours after administration of clopidogrel alone and in combination with LY2216684.
Time Frame: predose and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours postdose
Population: Participants with the CYP2C19*1/*1 genotype, who received at least 1 dose of clopidogrel, and had evaluable R-130964 plasma concentration data, including sufficient data in the terminal elimination phase for R-130964.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliters (h*ng/mL)
Groups:
- Clopidogrel: Clopidogrel: a single 300-milligram (mg) dose, administered orally on Day 1 of Treatment 1
- LY2216684 + Clopidogrel: LY2216684: 18-milligram (mg) dose, administered orally, once daily (QD) on Days 1 through 3 of Treatment 2
  Clopidogrel: a single 300-mg dose, administered orally on Day 3 of Treatment 2
Arm/Group | Clopidogrel | LY2216684 + Clopidogrel
Number analyzed (Participants) | 31 | 15
hours*nanograms/milliliters (h*ng/mL) | 61.8 (50) | 55.3 (44)

2. Primary Outcome: Pharmacokinetics of R-130964, Area Under the Concentration-time Curve From Time 0 to Time of Last Measurable Concentration (AUC0-tlast)
Description: R-130964 is the active metabolite of clopidogrel. Blood samples were collected prior to and through 24 hours after administration of clopidogrel alone and in combination with LY2216684. Log-transformed AUC0-tlast was analyzed using a linear mixed effects model with sequence, period, and treatment as fixed effects and participant as a random effect.
Time Frame: predose and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours postdose
Population: Participants with the CYP2C19*1/*1 genotype, who received at least 1 dose of clopidogrel, and had evaluable R-130964 plasma concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliters (h*ng/mL)
Arm/Group | Clopidogrel | LY2216684 + Clopidogrel
Number analyzed (Participants) | 38 | 36
hours*nanograms/milliliters (h*ng/mL) | 60.5 (45) | 46.9 (41)
Statistical Analysis 1: Comparison: Clopidogrel vs LY2216684 + Clopidogrel; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric Least Squares Means = 0.77, 90% CI 2-sided [0.72 to 0.83] — Statistical inference was made using the test treatment of LY2216684 + clopidogrel and the reference treatment of clopidogrel alone

3. Primary Outcome: Pharmacokinetics of R-130964, Maximum Observed Drug Concentrations (Cmax)
Description: R-130964 is the active metabolite of clopidogrel. Blood samples were collected prior to and through 24 hours after administration of clopidogrel alone and in combination with LY2216684. Log-transformed Cmax was analyzed using a linear mixed effects model with sequence, period, and treatment as fixed effects and participant as a random effect.
Time Frame: predose and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Clopidogrel | LY2216684 + Clopidogrel
Number analyzed (Participants) | 38 | 36
nanograms/milliliter (ng/mL) | 37.6 (56) | 22.7 (53)
Statistical Analysis 1: Comparison: Clopidogrel vs LY2216684 + Clopidogrel; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric Least Squares Means = 0.59, 90% CI 2-sided [0.53 to 0.67] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage Inhibition of Platelet Aggregation
Description: Blood samples for the measurement of platelet aggregation using a point-of-care device, Accumetrics VerifyNow™ P2Y12 (VN-P2Y12), were collected prior to and through 24 hours after administration of clopidogrel alone and in combination with LY2216684. Device-reported percent inhibition of VN-P2Y12 (IPRU) is presented.
Time Frame: predose and 2, 4, and 24 hours postdose
Population: Participants with the CYP2C19*1/*1 genotype, who received at least 1 dose of clopidogrel, and had evaluable IPRU data.
Measure: Mean (Standard Deviation); unit: IPRU
Arm/Group | Clopidogrel | LY2216684 + Clopidogrel
Number analyzed (Participants) | 38 | 37
IPRU
  Predose | 1.7 (3.2) | 1.4 (3.2)
  2 Hours Postdose | 16.0 (20.3) | 7.6 (12.3)
  4 Hours Postdose | 30.4 (21.8) | 14.0 (16.6)
  24 Hours Postdose | 25.1 (21.1) | 14.3 (17.5)

5. Primary Outcome: Pharmacokinetics of R-130964, Time to Maximum Observed Drug Concentrations (Tmax)
Description: as for outcome 1
Time Frame: predose and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Clopidogrel | LY2216684 + Clopidogrel
Number analyzed (Participants) | 36 | 36
hours | 1.50 [1.00 to 2.07] | 1.50 [0.50 to 4.00]
Statistical Analysis 1: Comparison: Clopidogrel vs LY2216684 + Clopidogrel; Test type: Superiority or Other; p = 0.3303, Wilcoxon (Mann-Whitney); Median of Paired Differences = 0.00, 90% CI 2-sided [0.00 to 0.25]

ADVERSE EVENTS:
Groups:
- Clopidogrel: Clopidogrel: a single 300-milligram (mg) dose, administered orally on Day 1
  Time Frame: Treatment 1
- LY2216684: LY2216684: 18-milligram (mg) dose, administered orally, once daily (QD) on Days 1 through 3
  Time Frame: Treatment 2; prior to clopidogrel dose on Day 3
- LY2216684 + Clopidogrel: LY2216684: 18-milligram (mg) dose, administered orally, once daily (QD) on Days 1 through 3
  Clopidogrel: a single 300-mg dose, administered orally on Day 3
  Time Frame: Treatment 2; after the clopidogrel dose on Day 3
Arm/Group | Clopidogrel | LY2216684 | LY2216684 + Clopidogrel
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 12/47 | 19/46 | 11/45
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel (N=47) | LY2216684 (N=46) | LY2216684 + Clopidogrel (N=45)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (8) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 2 (2)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 1 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (3)
Somnolence (Nervous system disorders) | 0 (0) | 7 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 4 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days